CLINICAL TRIAL: NCT05551559
Title: The Effect of Bariatric Surgery on Hepatic Metabolism in Non-Alcoholic Fatty Liver Disease
Acronym: BASIC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Panu Luukkonen, Adjunct Professor, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUS121992022
Record Dates: First submitted 2022-09-14; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Fatty Liver; Liver Diseases; Digestive System Diseases; Bariatric Surgery
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Liver Diseases; Digestive System Diseases | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bariatric surgery (Experimental)
  Interventions: Procedure: bariatric surgery

INTERVENTIONS:
Procedure: bariatric surgery — bariatric surgery

SUMMARY:
The purpose of this study is to investigate the mechanisms underlying bariatric surgery-induced resolution of non-alcoholic fatty liver disease.

DETAILED DESCRIPTION:
Bariatric surgery is one of the few currently available treatment options for non-alcoholic fatty liver disease (NAFLD). In most cases, NAFLD is entirely ameliorated after the surgery but in some individuals, the disease may persist or even progress. The mechanisms underlying the bariatric surgery-mediated resolution of NAFLD and the heterogeneity in the response remain poorly understood. In this study, the investigators will examine the metabolic effects of bariatric surgery-induced resolution of NAFLD. To this end, study subjects who have previously undergone bariatric surgery and metabolic studies will be invited for a follow-up visit for physical examination, evaluation of body composition with bioelectrical impedance and quantification of liver stiffness using non-invasive transient elastography and magnetic resonance elastography (MRE). Body fat composition will be evaluated by magnetic resonance imaging (MRI) and hepatic lipid content will be measured with magnetic resonance spectroscopy (MRS). In addition, 1H nuclear magnetic resonance (NMR) metabolomic analyses will be carried out from plasma samples collected both before and after bariatric surgery. Insulin resistance will be assessed using the HOMA-IR index and the genotypes in disease-modifying genes including PNPLA3, TM6SF2, MBOAT7, MARC1 and HSD17B13 will be assessed. Liver biopsies were obtained at the time of bariatric surgery and, in individuals with a clinical indication, a follow-up liver biopsy will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have undergone bariatric surgery and previously participated in a metabolic study in our research group.
* Participants must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
* Age range from 18-75 years.

Exclusion Criteria:

* No claustrophobia or metal implants to allow magnetic resonance spectroscopy.
* No pregnancy or lactation in women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
change in concentration of plasma metabolites as determined by nuclear magnetic resonance | change between follow-up visit and pre-surgery visit , expected average 10 years
  plasma NMR metabolomics concentrations (mmol/L)
change in severity of NAFLD as determined by elastography | change between follow-up visit and pre-surgery visit , expected average 10 years
  elastography (kPa)
change in severity of NAFLD as determined by magnetic resonance spectroscopy | change between follow-up visit and pre-surgery visit , expected average 10 years
  intrahepatic triglyceride content by proton magnetic resonance spectroscopy (%)
change in severity of NAFLD as determined by liver histology | change between follow-up visit and pre-surgery visit , expected average 10 years
  liver biopsy from individuals with clinical indication (SAF score)

CONTACTS AND LOCATIONS:
Overall Officials: Panu K Luukkonen, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Biomedicum 2U, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No